CLINICAL TRIAL: NCT05687214
Title: Investigation on the Effects of an Osteopathic Manipulative Treatment for Constipation in People With Rett Syndrome
Brief Title: Osteopathic Manipulative Treatment for Constipation in People With Rett Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Collaborators: Associazione Italiana Rett (AIRETT) (Unknown)
Responsible Party: Principal Investigator, Meir Lotan, Professor, Ariel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AU-HEA-ML-20220915
Record Dates: First submitted 2022-12-30; First posted 2023-01-18 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Single-blind parallel group-randomized design.
Who Masked: Outcomes Assessor
Masking Description: The assessors will not know which group the participants were assigned (experimental or control group) at any study stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each participant in the experimental group will receive eight weekly osteopathic manipulative treatments within eight weeks. Each treatment session will include several specific manipulations.
  Interventions: Other: Osteopathic manipulative treatment
- Control Group (No Intervention): Participants in the control group will not receive any treatment.

INTERVENTIONS:
Other: Osteopathic manipulative treatment — Each participant in the experimental group will receive eight osteopathic manipulative treatments. Each treatment will include the following manipulations:
  * Pompage Cv4;
  * Occipital-sternal technique;
  * Relaxining manipulation of the diaphragmatic domes;
  * Pelvic and abdominal diaphragm synchronization;
  * Dynamogenic technique;
  * Mesenteric traction;
  * Release of colic angles;
  * Manipulation and mobilization of the sacrum.
  Arms: Experimental group

SUMMARY:
Constipation consists of bowel symptoms characterized by difficulty or infrequency passage of stool, stiff stool, or a feeling of incomplete evacuation. However, its impact goes far beyond this definition. Constipation negatively impacts the quality of life (QoL) of children and adults suffering from this condition, affecting mental and physical-related QoL. Additionally, a negative impact of constipation on QoL was found in parents carrying children with constipation, affecting family functioning.

People with an intellectual disability present a constipation rate of over 33%. Rett syndrome (RTT) is a complex neurodevelopmental disorder affecting about 1/10,000 females and a few males worldwide. Chronic constipation is persistent in people with RTT, with a reported prevalence higher than 74%.

Specific recommendations for constipation management in RTT were developed, including behavioral, pharmacological, and surgical considerations. Recently, the literature has been enriched with papers describing the osteopathic treatment efficacy in reducing constipation. Emerging literature reported the efficacy of OMT in reducing constipation symptoms and improving QoL in typically developed people, as well as in children with disability. The present study aims to evaluate the efficacy of a specific OMT for managing chronic constipation in people with RTT and its impact on primary caregivers' quality of life.

Research questions:

* Can an OMT improve the constipation of people with RTT, increasing the frequency of bowel movements?
* Can the effects of an OMT aimed at reducing the constipation symptoms in people with RTT positively impact the participants' parents' constipation-related QoL?

Twelve individuals with RTT and their families will be recruited to participate in this single-blind parallel group-randomized study. Participants will be randomly divided into an experimental group (EG) and a control group (CG). After the preliminary evaluations, each participant will undergo eight OMT carried out weekly for eight weeks. The OMT will aim to facilitate bowel movements by increasing blood flow through the abdomen. At the end of the treatment, the participants will repeat the evaluation conducted before the OMT, and the collected data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of classic Rett syndrome with a mutation of the MECP2 gene;
* matching the ROME IV criteria for constipation;

Exclusion Criteria:

* the presence of specific severe heart and cardiovascular diseases;
* the presence of amenorrhea.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Change in number of evacuations | Every day, for one week, immediately before the intervention phase.
  The number of participants' evacuations collected daily by participants' caregivers
Change in number of evacuations | Every day, during the intervention phase (for 8 weeks).
  The number of participants' evacuations collected daily by participants' caregivers
Change in number of evacuations | Every day, for one week, immediately after the end of the intervention phase.
  The number of participants' evacuations collected daily by participants' caregivers
Change in number of enemas and medications | Every day, for one week, immediately before the intervention phase.
  The number of enemas and medication provided to the participants' to simplify or induce the evacuations collected by their caregivers.
Change in number of enemas and medications | Every day, during the intervention phase (for 8 weeks).
  The number of enemas and medication provided to the participants' to simplify or induce the evacuations collected by their caregivers.
Change in number of enemas and medications | Every day, for one week, immediately after the end of the intervention phase.
  The number of enemas and medication provided to the participants' to simplify or induce the evacuations collected by their caregivers.
Change in the Modified Constipation Assessment Scale (m-CAS) | 15 minutes. Before the treatment initiation (T0) and after the treatment end (T1 - after 8 weeks from T0).
  The m-CAS is an eight-item scale that measures whether constipation is present and its intensity. A higher score represents more severe constipation. Cronbach α coefficient showed good internal consistency over time (α>0.70). The Pearson product-moment correlation coefficient was used to evaluate test-retest reliability and showed evident acceptance (r=0.93; P<0.001).
Change in theConstipation Scoring System (CSS) | 15 minutes. Before the treatment initiation (T0) and after the treatment end (T1 - after 8 weeks from T0).
  The CSS assesses the severity of constipation with a maximum score of 30 (0 = no constipation, 30 = severe constipation. The scale was initially validated with a 100-subject sample and could correctly detect the absence or presence of constipation in 96% of the subjects, thus representing a sensitive and valid tool.
Change in theConstipation-Related Quality Of Life (CRQOL) | 15 minutes. Before the treatment initiation (T0) and after the treatment end (T1 - after 8 weeks from T0).
  The CRQOL assesses quality-of-life domains affected by constipation. It includes four domains: social impairment, distress, eating habits, and bathroom attitudes. In our study, the primary caregiver filled this scale reporting his feelings concerning the participant's constipation management. The internal consistency of each of the four domains was higher than 0.70 using Cronbach's alpha. Excellent test-retest reliability was demonstrated (α>0.85).
Change in the Short Form Health Survey-12 (SF-12) | 15 minutes. Before the treatment initiation (T0) and after the treatment end (T1 - after 8 weeks from T0).
  The SF-12 is a multidimensional measure of health-related quality of life widely used in clinical trials. The SF-12 was administered to participants' primary caregivers. The Italian version of the SF-12 was validated on a large sample of Italian people showing strong psychometric proprieties.

SECONDARY OUTCOMES:
Change in the tissue tension | 15 minutes. Before the treatment initiation (T0) and after the treatment end (T1 - after 8 weeks from T0).
  The pelvic tissue tension was evaluated as an index of hydration and deep fascial tension. For the assessment, the iliac cavity skin was pinched between the index and thumb fingers, and a score between 0 (normal tissue elasticity) and 4 (adherent, rigid skin, tissue detachment not possible) was assigned based on the tissue elasticity.
Change in the abdomen palpability | 15 minutes. Before the treatment initiation (T0) and after the treatment end (T1 - after 8 weeks from T0).
  It represents an index of abdominal stiffness and refers to the intestinal skein resistance to manual mobilization in the supine position. The right and left colic cords, ileocecal valve, and sigma were mobilized. Based on the perceived tissue consistency and resistance, scores between 0 (soft and treatable abdominal tissue) and 3 (rigid abdomen, tense and painful even in the medium-deep palpation) points were assigned.
Change in the abdominal bloating | 15 minutes. Before the treatment initiation (T0) and after the treatment end (T1 - after 8 weeks from T0).
  It assesses the presence and extent of intestinal gas. It is helpful to have an approximate idea of the intestinal loops' opening (or closing) level. It was assessed by observing the prominence of the four abdominal quadrants in correspondence with the navel, anterior iliac thorns, and costal ramps. And a score between 0 (flat, compressible abdomen) and 4 (globose abdomen, total compressibility not possible) was assigned.
Change in the sacral pad swelling | 15 minutes. Before the treatment initiation (T0) and after the treatment end (T1 - after 8 weeks from T0).
  Its presence can indicate inadequate liquids' reabsorption in the small pelvis by the iliac branches. It is evaluated in the supine position by manual pressure examination of the sacral base. Based on the sacral area swelling, a score between 0 (normally distended sacral area) and 3 (large swelling with lumbar-sacral area tissue inhibition).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Angela Fabio, PhD, Principal Investigator — Department of Clinical and Experimental Medicine, University of Messina
Locations (1):
- Centro AIRETT Ricerca e Innovazione (CARI), Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the anonymized IPD related to participants' age, and levels of Rett syndrome severity, motor functioning, and daily physical activity. The information will be published as a part of the scientific articles produced after the study ends.
Time Frame: The IPD will be available if and when scientific articles related to this study are published. Should the data be published, they will be available indefinitely in the scientific literature.
Access Criteria: The investigators plan to submit scientific articles related to the present study to be published in an open access peer-review scientific journal. Therefore, if the articles are published, the data will be available on the website of the journal in which they were published.

REFERENCES:
- [Background] Bharucha AE, Pemberton JH, Locke GR 3rd. American Gastroenterological Association technical review on constipation. Gastroenterology. 2013 Jan;144(1):218-38. doi: 10.1053/j.gastro.2012.10.028. No abstract available. PMID 23261065
- [Background] Sbahi H, Cash BD. Chronic Constipation: a Review of Current Literature. Curr Gastroenterol Rep. 2015 Dec;17(12):47. doi: 10.1007/s11894-015-0471-z. PMID 26449614
- [Background] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Background] Jani B, Marsicano E. Constipation: Evaluation and Management. Mo Med. 2018 May-Jun;115(3):236-240. PMID 30228729
- [Background] Leung L, Riutta T, Kotecha J, Rosser W. Chronic constipation: an evidence-based review. J Am Board Fam Med. 2011 Jul-Aug;24(4):436-51. doi: 10.3122/jabfm.2011.04.100272. PMID 21737769
- [Background] Vriesman MH, Rajindrajith S, Koppen IJN, van Etten-Jamaludin FS, van Dijk M, Devanarayana NM, Tabbers MM, Benninga MA. Quality of Life in Children with Functional Constipation: A Systematic Review and Meta-Analysis. J Pediatr. 2019 Nov;214:141-150. doi: 10.1016/j.jpeds.2019.06.059. Epub 2019 Aug 6. PMID 31399248
- [Background] Wang C, Shang L, Zhang Y, Tian J, Wang B, Yang X, Sun L, Du C, Jiang X, Xu Y. Impact of functional constipation on health-related quality of life in preschool children and their families in Xi'an, China. PLoS One. 2013 Oct 10;8(10):e77273. doi: 10.1371/journal.pone.0077273. eCollection 2013. PMID 24130872
- [Background] Kaugars AS, Silverman A, Kinservik M, Heinze S, Reinemann L, Sander M, Schneider B, Sood M. Families' perspectives on the effect of constipation and fecal incontinence on quality of life. J Pediatr Gastroenterol Nutr. 2010 Dec;51(6):747-52. doi: 10.1097/MPG.0b013e3181de0651. PMID 20706148
- [Background] Thompson AP, MacDonald SE, Wine E, Scott SD. Understanding Parents' Experiences When Caring for a Child With Functional Constipation: Interpretive Description Study. JMIR Pediatr Parent. 2021 Jan 20;4(1):e24851. doi: 10.2196/24851. PMID 33470939
- [Background] De Hert M, Hudyana H, Dockx L, Bernagie C, Sweers K, Tack J, Leucht S, Peuskens J. Second-generation antipsychotics and constipation: a review of the literature. Eur Psychiatry. 2011 Jan;26(1):34-44. doi: 10.1016/j.eurpsy.2010.03.003. Epub 2010 Jun 9. PMID 20542667
- [Background] Balogh RS, Ouellette-Kuntz H, Brownell M, Colantonio A. Ambulatory Care Sensitive Conditions in Persons with an Intellectual Disability - Development of a Consensus. J Appl Res Intellect Disabil 2011;24:150-8. doi:10.1111/j.1468-3148.2010.00578.x.
- [Background] Bosch J, Van Dyke C, Smith SM, Poulton S. Role of medical conditions in the exacerbation of self-injurious behavior: an exploratory study. Ment Retard. 1997 Apr;35(2):124-30. doi: 10.1352/0047-6765(1997)0352.0.CO;2. PMID 9131872
- [Background] Carr EG, Smith CE. Biological setting events for self-injury. Ment Retard Dev Disabil Res Rev 1995;1:94-8. doi:10.1002/mrdd.1410010204.
- [Background] Christensen TJ, Ringdahl JE, Bosch JJ, Falcomata TS, Luke JR, Andelman MS. Constipation associated with self-injurious and aggressive behavior exhibited by a child diagnosed with autism. Educ Treat Child 2009;32:89-103. doi:10.1353/etc.0.0041.
- [Background] Coleman J, Spurling G. Constipation in people with learning disability. BMJ. 2010 Jan 26;340:c222. doi: 10.1136/bmj.c222. No abstract available. PMID 20103526
- [Background] Robertson J, Chadwick D, Baines S, Emerson E, Hatton C. Prevalence of Dysphagia in People With Intellectual Disability: A Systematic Review. Intellect Dev Disabil. 2017 Dec;55(6):377-391. doi: 10.1352/1934-9556-55.6.377. PMID 29194030
- [Background] Fombonne E, Simmons H, Ford T, Meltzer H, Goodman R. Prevalence of pervasive developmental disorders in the British nationwide survey of child mental health. Int Rev Psychiatry. 2003 Feb-May;15(1-2):158-65. doi: 10.1080/0954026021000046119. PMID 12745327
- [Background] Skjeldal OH, von Tetzchner S, Aspelund F, Herder GA, Lofterld B. Rett syndrome: geographic variation in prevalence in Norway. Brain Dev. 1997 Jun;19(4):258-61. doi: 10.1016/s0387-7604(97)00572-x. PMID 9187475
- [Background] Pini G, Milan M, Zappella M. Rett syndrome in northern Tuscany (Italy): family tree studies. Clin Genet. 1996 Dec;50(6):486-90. doi: 10.1111/j.1399-0004.1996.tb02718.x. PMID 9147879
- [Background] Amir RE, Van den Veyver IB, Wan M, Tran CQ, Francke U, Zoghbi HY. Rett syndrome is caused by mutations in X-linked MECP2, encoding methyl-CpG-binding protein 2. Nat Genet. 1999 Oct;23(2):185-8. doi: 10.1038/13810. PMID 10508514
- [Background] Neul JL, Kaufmann WE, Glaze DG, Christodoulou J, Clarke AJ, Bahi-Buisson N, Leonard H, Bailey ME, Schanen NC, Zappella M, Renieri A, Huppke P, Percy AK; RettSearch Consortium. Rett syndrome: revised diagnostic criteria and nomenclature. Ann Neurol. 2010 Dec;68(6):944-50. doi: 10.1002/ana.22124. PMID 21154482
- [Background] Epstein LG. Rett Syndrome--Clinical and Biological Aspects: Studies on 130 Swedish Females. Arch Neurol 1995;52:343-4. doi:10.1001/archneur.1995.00540280025011.
- [Background] Hagberg B, Aicardi J, Dias K, Ramos O. A progressive syndrome of autism, dementia, ataxia, and loss of purposeful hand use in girls: Rett's syndrome: report of 35 cases. Ann Neurol. 1983 Oct;14(4):471-9. doi: 10.1002/ana.410140412. PMID 6638958
- [Background] Hagberg B, Anvret M, Wahlstrom J, Wahlström J. Rett syndrome-Clinical and biological aspects: Studies on 130 Swedish females. London: Cambridge University Press; 1993.
- [Background] Hagberg B. Clinical manifestations and stages of Rett syndrome. Ment Retard Dev Disabil Res Rev. 2002;8(2):61-5. doi: 10.1002/mrdd.10020. PMID 12112728
- [Background] Schwartzman F, Vitolo MR, Schwartzman JS, Morais MB. Eating practices, nutritional status and constipation in patients with Rett syndrome. Arq Gastroenterol. 2008 Oct-Dec;45(4):284-9. doi: 10.1590/s0004-28032008000400005. English, Portuguese. PMID 19148355
- [Background] Strati F, Cavalieri D, Albanese D, De Felice C, Donati C, Hayek J, Jousson O, Leoncini S, Pindo M, Renzi D, Rizzetto L, Stefanini I, Calabro A, De Filippo C. Altered gut microbiota in Rett syndrome. Microbiome. 2016 Jul 30;4(1):41. doi: 10.1186/s40168-016-0185-y. PMID 27473171
- [Background] Morton RE, Bonas R, Minford J, Kerr A, Ellis RE. Feeding ability in Rett syndrome. Dev Med Child Neurol. 1997 May;39(5):331-5. doi: 10.1111/j.1469-8749.1997.tb07440.x. PMID 9236700
- [Background] Motil KJ, Schultz RJ, Browning K, Trautwein L, Glaze DG. Oropharyngeal dysfunction and gastroesophageal dysmotility are present in girls and women with Rett syndrome. J Pediatr Gastroenterol Nutr. 1999 Jul;29(1):31-7. doi: 10.1097/00005176-199907000-00010. PMID 10400100
- [Background] Schultz RJ, Glaze DG, Motil KJ, Armstrong DD, del Junco DJ, Hubbard CR, Percy AK. The pattern of growth failure in Rett syndrome. Am J Dis Child. 1993 Jun;147(6):633-7. doi: 10.1001/archpedi.1993.02160300039018. PMID 8506830
- [Background] Tsiropoulos I, Andersen M, Hallas J. Adverse events with use of antiepileptic drugs: a prescription and event symmetry analysis. Pharmacoepidemiol Drug Saf. 2009 Jun;18(6):483-91. doi: 10.1002/pds.1736. PMID 19326363
- [Background] Every-Palmer S, Newton-Howes G, Clarke MJ. Pharmacological treatment for antipsychotic-related constipation. Cochrane Database Syst Rev. 2017 Jan 24;1(1):CD011128. doi: 10.1002/14651858.CD011128.pub2. PMID 28116777
- [Background] Romano A, Di Rosa G, Tisano A, Fabio RA, Lotan M. Effects of a remotely supervised motor rehabilitation program for individuals with Rett syndrome at home. Disabil Rehabil. 2022 Oct;44(20):5898-5908. doi: 10.1080/09638288.2021.1949398. Epub 2021 Jul 20. PMID 34282992
- [Background] Percy AK, Lee HS, Neul JL, Lane JB, Skinner SA, Geerts SP, Annese F, Graham J, McNair L, Motil KJ, Barrish JO, Glaze DG. Profiling scoliosis in Rett syndrome. Pediatr Res. 2010 Apr;67(4):435-9. doi: 10.1203/PDR.0b013e3181d0187f. PMID 20032810
- [Background] Romano A, Ippolito E, Risoli C, Malerba E, Favetta M, Sancesario A, Lotan M, Moran DS. Intensive Postural and Motor Activity Program Reduces Scoliosis Progression in People with Rett Syndrome. J Clin Med. 2022 Jan 22;11(3):559. doi: 10.3390/jcm11030559. PMID 35160011
- [Background] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575
- [Background] Baikie G, Ravikumara M, Downs J, Naseem N, Wong K, Percy A, Lane J, Weiss B, Ellaway C, Bathgate K, Leonard H. Gastrointestinal dysmotility in Rett syndrome. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):237-44. doi: 10.1097/MPG.0000000000000200. PMID 24121144
- [Background] Budden SS. Management of Rett syndrome: a ten year experience. Neuropediatrics. 1995 Apr;26(2):75-7. doi: 10.1055/s-2007-979727. PMID 7566457
- [Background] Tse PW, Leung SS, Chan T, Sien A, Chan AK. Dietary fibre intake and constipation in children with severe developmental disabilities. J Paediatr Child Health. 2000 Jun;36(3):236-9. doi: 10.1046/j.1440-1754.2000.00498.x. PMID 10849223
- [Background] Tolia V, Ventimiglia J, Kuhns L. Gastrointestinal tolerance of a pediatric fiber formula in developmentally disabled children. J Am Coll Nutr. 1997 Jun;16(3):224-8. doi: 10.1080/07315724.1997.10718678. PMID 9176828
- [Background] Bosch, J.; Mraz, R.; Masbruch, J.; Tabor, A.; Van Dyke, D.; McBrien, D. Constipation in Young Children with Developmental Disabilities. Infants Young Child 2002, 15, 66-77, doi:10.1097/00001163-200210000-00009.
- [Background] American College of Gastroenterology Chronic Constipation Task Force. An evidence-based approach to the management of chronic constipation in North America. Am J Gastroenterol. 2005;100 Suppl 1:S1-4. doi: 10.1111/j.1572-0241.2005.50613_1.x. No abstract available. PMID 16008640
- [Background] Matson JL, LoVullo SV. Encopresis, soiling and constipation in children and adults with developmental disability. Res Dev Disabil. 2009 Jul-Aug;30(4):799-807. doi: 10.1016/j.ridd.2008.12.001. Epub 2009 Jan 21. PMID 19162439
- [Background] Ternent CA, Bastawrous AL, Morin NA, Ellis CN, Hyman NH, Buie WD; Standards Practice Task Force of The American Society of Colon and Rectal Surgeons. Practice parameters for the evaluation and management of constipation. Dis Colon Rectum. 2007 Dec;50(12):2013-22. doi: 10.1007/s10350-007-9000-y. No abstract available. PMID 17665250
- [Background] Constipation Guideline Committee of the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. Evaluation and treatment of constipation in infants and children: recommendations of the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. J Pediatr Gastroenterol Nutr. 2006 Sep;43(3):e1-13. doi: 10.1097/01.mpg.0000233159.97667.c3. PMID 16954945
- [Background] Hundscheid HW, Pepels MJ, Engels LG, Loffeld RJ. Treatment of irritable bowel syndrome with osteopathy: results of a randomized controlled pilot study. J Gastroenterol Hepatol. 2007 Sep;22(9):1394-8. doi: 10.1111/j.1440-1746.2006.04741.x. PMID 17716344
- [Background] Tarsuslu T, Bol H, Simsek IE, Toylan IE, Cam S. The effects of osteopathic treatment on constipation in children with cerebral palsy: a pilot study. J Manipulative Physiol Ther. 2009 Oct;32(8):648-53. doi: 10.1016/j.jmpt.2009.08.016. PMID 19836601
- [Background] Fernandes WVB, Blanco CR, Politti F, de Cordoba Lanza F, Lucareli PRG, Correa JCF. The effect of a six-week osteopathic visceral manipulation in patients with non-specific chronic low back pain and functional constipation: study protocol for a randomized controlled trial. Trials. 2018 Mar 2;19(1):151. doi: 10.1186/s13063-018-2532-8. PMID 29499728
- [Background] Brugman, R.; Fitzgerald, K.; Fryer, G. The Effect of Osteopathic Treatment on Chronic Constipation - A Pilot Study. International Journal of Osteopathic Medicine 2010, 13, 17-23, doi:10.1016/j.ijosm.2009.10.002.
- [Background] Belvaux A, Bouchoucha M, Benamouzig R. Osteopathic management of chronic constipation in women patients. Results of a pilot study. Clin Res Hepatol Gastroenterol. 2017 Oct;41(5):602-611. doi: 10.1016/j.clinre.2016.12.003. Epub 2017 Feb 16. PMID 28215390
- [Background] Zollars JA, Armstrong M, Whisler S, Williamson S. Visceral and Neural Manipulation in Children with Cerebral Palsy and Chronic Constipation: Five Case Reports. Explore (NY). 2019 Jan-Feb;15(1):47-54. doi: 10.1016/j.explore.2018.09.001. Epub 2018 Sep 6. PMID 30528865
- [Background] Smith, L.; Berkowitz, M.R. Osteopathic Approach to Chronic Constipation in Prader-Willi Syndrome: A Case Report. International Journal of Osteopathic Medicine 2016, 19, 73-77, doi:10.1016/J.IJOSM.2015.11.002.
- [Background] Aquino A, Perini M, Cosmai S, Zanon S, Pisa V, Castagna C, Uberti S. Osteopathic Manipulative Treatment Limits Chronic Constipation in a Child with Pitt-Hopkins Syndrome. Case Rep Pediatr. 2017;2017:5437830. doi: 10.1155/2017/5437830. Epub 2017 Jan 31. PMID 28251008
- [Background] Rodocanachi Roidi ML, Isaias IU, Cozzi F, Grange F, Scotti FM, Gestra VF, Gandini A, Ripamonti E. A New Scale to Evaluate Motor Function in Rett Syndrome: Validation and Psychometric Properties. Pediatr Neurol. 2019 Nov;100:80-86. doi: 10.1016/j.pediatrneurol.2019.03.005. Epub 2019 Mar 16. PMID 31047758
- [Background] Romano A, Capri T, Semino M, Bizzego I, Di Rosa G, Fabio RA. Gross Motor, Physical Activity and Musculoskeletal Disorder Evaluation Tools for Rett Syndrome: A Systematic Review. Dev Neurorehabil. 2020 Nov;23(8):485-501. doi: 10.1080/17518423.2019.1680761. Epub 2019 Oct 31. PMID 31668104
- [Background] Lor L, Hill K, Jacoby P, Leonard H, Downs J. A validation study of a modified Bouchard activity record that extends the concept of 'uptime' to Rett syndrome. Dev Med Child Neurol. 2015 Dec;57(12):1137-42. doi: 10.1111/dmcn.12838. Epub 2015 Jun 23. PMID 26108439
- [Background] Fabio, R.A.; Martinazzoli, C.; Antonietti, A. Development and Standardization of the "Rars"(Rett Assessment Rating Scale). Life Span Disabil 2005, 8, 257-281.
- [Background] Woolery M, Carroll E, Fenn E, Wieland H, Jarosinski P, Corey B, Wallen GR. A constipation assessment scale for use in pediatric oncology. J Pediatr Oncol Nurs. 2006 Mar-Apr;23(2):65-74. doi: 10.1177/1043454205285874. PMID 16476780
- [Background] Agachan F, Chen T, Pfeifer J, Reissman P, Wexner SD. A constipation scoring system to simplify evaluation and management of constipated patients. Dis Colon Rectum. 1996 Jun;39(6):681-5. doi: 10.1007/BF02056950. PMID 8646957
- [Background] Wang JY, Hart SL, Lee J, Berian JR, McCrea GL, Varma MG. A valid and reliable measure of constipation-related quality of life. Dis Colon Rectum. 2009 Aug;52(8):1434-42. doi: 10.1007/DCR.0b013e3181a51196. PMID 19617757
- [Background] Kodraliu G, Mosconi P, Groth N, Carmosino G, Perilli A, Gianicolo EA, Rossi C, Apolone G. Subjective health status assessment: evaluation of the Italian version of the SF-12 Health Survey. Results from the MiOS Project. J Epidemiol Biostat. 2001;6(3):305-16. doi: 10.1080/135952201317080715. PMID 11437095
- [Background] Curi ACC, Maior Alves AS, Silva JG. Cardiac autonomic response after cranial technique of the fourth ventricle (cv4) compression in systemic hypertensive subjects. J Bodyw Mov Ther. 2018 Jul;22(3):666-672. doi: 10.1016/j.jbmt.2017.11.013. Epub 2017 Dec 9. PMID 30100295
- [Background] Milnes, K.; Moran, R.W. Physiological Effects of a CV4 Cranial Osteopathic Technique on Autonomic Nervous System Function: A Preliminary Investigation. International Journal of Osteopathic Medicine 2007, 10, 8-17, doi:10.1016/j.ijosm.2007.01.003.
- [Background] Paoletti, S. Le Fasce: Il Ruolo Dei Tessuti Nella Meccanica Umana; ESOMM: Rome, IT, 2003; ISBN 0157347362.
- [Background] Barral, J.P. Advanced Visceral Manipulation: Neuroendocrine Approach to the Abdomen; The Barral Institute: Ayr, UK, 2020; ISBN 9780998747965.
- [Background] Bordoni, B.D. I Cinque Diaframmi. Medicina Manuale; Edi.Ermes: Milano, IT, 2021; ISBN 9788870517415.
- [Background] Weischenck, J. Traité d Ostéopathie Viscérale; Maloine S.A.: Paris, FR, 1982; ISBN 9788874490929.
- [Background] American Osteopathic Association Foundations of Osteopathic Medicine; Chila, A.G., Carreiro, J.E., Dowling, D.J., Gamber, R.G., Glover, J.C., Habenicht, A.L., Jerome, J.A., Patterson, M.M., Rogers, F.J., Seffinger, M.A., Willard, F.H., Eds.; 3rd ed.; Lippincott Williams & Wilkins: Philadelphia, PA, 2015; ISBN 9780781766715.
- [Background] Kapandji, I.A. The Physiology of the Joints: The Spinal Column, Pelvic Girdle and Head; 7th ed.; Handspring Publishing: London, UK, 2019; ISBN 9781912085613.